CLINICAL TRIAL: NCT03967561
Title: Effects of Progressive vs. Non-progressive Water-based Aerobic Training on Type 2 Diabetes Control: a Randomized Clinical Trial
Brief Title: Progressive vs. Non-progressive Water-based Aerobic Training on Type 2 Diabetes Control: a Randomized Clinical Trial
Acronym: PAT-DM2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Luiz Fernando Martins Kruel, Associate professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2.855.513
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Exercise; Water-based exercise; Aerobic exercise; Glucose control; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial with two interventions in parallel.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive aerobic training (Experimental): Water-based aerobic training performed with progression in the training variables. The intervention will be performed during 12 weeks, with 3 weekly sessions (of 50 minutes each), of walking/running in shallow pool.
  Interventions: Other: Progressive water-based aerobic training
- Non-progressive aerobic training (Experimental): Water-based aerobic training performed without progression in the training variables. The intervention will be performed during 12 weeks, with 3 weekly sessions (of 50 minutes each), of walking/running in shallow pool.
  Interventions: Other: Non-progressive aerobic training

INTERVENTIONS:
Other: Progressive water-based aerobic training — The intervention will comprise walking/running in shallow pool with progression in the training variables. The training will have 12 weeks of duration with 3 weekly sessions (of 50 minutes each).
  Arms: Progressive aerobic training
Other: Non-progressive aerobic training — The intervention will comprise walking/running in shallow pool without progression in the training variables. The training will have 12 weeks of duration with 3 weekly sessions (of 50 minutes each).
  Arms: Non-progressive aerobic training

SUMMARY:
This is a randomized clinical trial with the aim to evaluate the effects of two water-based aerobic training programs (walking or running in shallow pool) on type 2 diabetes control. The sample will be composed by 50 individuals with type 2 diabetes, of both sexes, aged between 40 and 70 years, who will be randomized into water-based progressive aerobic training (PAT, n=25) and water-based non-progressive aerobic training (NPAT, n=25). Both trainings will have 12 weeks of duration with 3 weekly sessions (of 50 minutes each). Biochemical, cardiorespiratory fitness, maximum strength, body composition and functional mobility variables, as also quality of life, sleep quality and depressive symptoms will be analyzed before and after the 12 weeks of training.

DETAILED DESCRIPTION:
Water-based aerobic training can provide benefits with important clinical implications for type 2 diabetes (T2D) patients, as the aquatic environment provides some interesting advantages to this population. The lower impact on joints and consequent reduced chance of injury allows considering the aquatic environment favorable to the principle of continuity with progression of physiological stimuli and metabolic benefits.

In T2D individuals, studies have been analyzing the effects of water-based aerobic training in upright position, which have been promoting several results in metabolic parameters of T2D individuals, including benefits in glucose and lipids levels and in cardiorespiratory fitness.

The literature shows distinct exercise effects on glucose control of T2D patients, resulting from different forms of training structuring, with and without progression of training variables. Well-conducted clinical trials prescribing aerobic training according to American Diabetes Association (ADA) recommendations (i.e. structured aerobic training with weekly duration of at least 150 minutes of moderate to vigorous intensity performed in three or more sessions per week) but with minimal or without progression in training load found no HbA1c reductions, whereas some studies that did not meet the recommendations but progressed training volume and/or intensity over time found interesting HbA1c reductions. With these findings, it seems that the optimization of aerobic training benefits on glucose control may not solely depend on a fixed training dosage, but also on the progression of the volume and/or intensity of training.

Due to the associations between T2D with obesity and hypertension, conditions that create difficulties for individuals performing exercise while supporting their own body mass, the different responses arising from the studies investigating progressive and non-progressive aerobic trainings in T2D patients, and with the important facilities that the aquatic environment can promote during physical exercise performance, it becomes interesting to investigate the effects of the application of two aquatic aerobic trainings on T2D treatment, in which similar exercise programs are performed, with one of them having its training variables fixed over time (non-progressive training) and the other with progression in the variables (progressive training). To the present moment, no clinical trial has investigated the comparison between aquatic aerobic training interventions with and without progression in the training variables on glycemic control of T2D individuals, aiming at exploring the role of training progression.

For this purpose, a randomized clinical trial with the aim to evaluate the effects of two water-based aerobic training programs (walking or running in shallow pool) on T2D management will be performed. The sample will be composed by 50 individuals with T2D, of both sexes, aged between 40 and 70 years, who will be randomized into water-based progressive aeroibic training (PAT, n=25) and water-based non-progressive aerobic training (NPAT, n=25). Both trainings will have 12 weeks of duration with 3 weekly sessions (of 50 minutes each). Biochemical, cardiorespiratory fitness, maximum strength, body composition and functional mobility variables, as also quality of life, sleep quality and depressive symptoms will be analyzed before and after the 12 weeks of training.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with type 2 diabetes, of both sexes, aged between 40 and 70 years.
* Be under medical treatment with oral hypoglycemic agents and / or insulin;
* Not be engaged in regular exercise (regular exercise was defined as performing any type of physical training for at least 20 minutes three or more days a week).

Exclusion Criteria:

* Presence of:
* uncontrolled hypertension;
* autonomic neuropathy;
* severe peripheral neuropathy;
* proliferative diabetic retinopathy;
* severe non-proliferative diabetic retinopathy;
* uncompensated heart failure;
* peripheral amputations;
* chronic kidney failure;
* body mass index (BMI)> 45.0 kg/m2;
* to have some muscle or joint impairment that prevents the performance of physical exercises safely.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-06-10 (Estimated); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-11-15 (Estimated)

PRIMARY OUTCOMES:
Glycated Hemoglobin levels (HbA1c) | Change from baseline levels of glycated hemoglobin to 12 weeks of intervention.
  Blood samples will be used to analyze glycated hemoglobin levels (%)

SECONDARY OUTCOMES:
Fasting plasma glucose | At baseline and after a 12-week period
  in mg/dL
Fasting insulin | At baseline and after a 12-week period
  in mg/dL
Insulin-resistance index (HOMA-IR) | At baseline and after a 12-week period
  in amount
Total cholesterol | At baseline and after a 12-week period
  in mg/dL
High density lipoprotein | At baseline and after a 12-week period
  in mg/dL
Low density lipoprotein | At baseline and after a 12-week period
  in mg/dL
Triglycerides | At baseline and after a 12-week period
  in mg/dL
Plasma renin | At baseline and after a 12-week period
  in uIU/mL (microliter)
C-reactive protein | At baseline and after a 12-week period
  in mg/L
Peak oxygen uptake | At baseline and after a 12-week period
  in ml.kg.min-1
Oxygen uptake at the second ventilatory threshold. | At baseline and after a 12-week period
  in ml.kg.min-1
Percentage of oxygen consumption in the second ventilatory threshold from the peak oxygen uptake | At baseline and after a 12-week period
  in %
Systolic blood pressure. | At baseline and after a 12-week period
  in mmHg
Diastolic blood pressure. | At baseline and after a 12-week period
  in mmHg
Resting heart rate | At baseline and after a 12-week period
  in beats per minute
Maximum dynamic muscle strength (1RM) in the knees extension exercise | At baseline and after a 12-week period
  The test is characterized by greatest load that can be supported in a single execution of knees extension exercise.
Muscular resistance (maximal repetitions) in the knees extension exercise. | At baseline and after a 12-week period
  To determine muscular resistance, it will be considered the number of repetitions performed at 60% of 1RM, following a paced pre-established execution. In the post-training evaluation, we will use the load of 60% of 1RM test performed in the pre-training.
Timed up-and-go test performed at the usual speed. | At baseline and after a 12-week period
  In seconds
Timed up-and-go test performed at the maximal speed. | At baseline and after a 12-week period
  In seconds
Overall quality of life and in physical, psychological, social relationships and environment domains, evaluated by instrument of World Health Organization (WHOQOL). | At baseline and after a 12-week period
  To evaluate the quality of life we used the WHOQOL-brief instrument. This instrument is self-applicable, cross-cultural, translated and validated for Portuguese, consisting of 26 questions. Its score ranges from zero to 100 points, divided into the physical, psychological, social relationships and environment, as well as an assessment of the overall quality of life.
Depressive symptoms, evaluated by Depression Inventory Patient Health Questionnaire (PHQ-9) | At baseline and after a 12-week period
  For evaluation of depressive symptoms was used the questionnaire PHQ-9 depression, which consists of nine items, including symptoms and attitudes whose intensity varies from zero to three, with 27 being the higher score.
Sleep quality, evaluated by Pittsburgh Sleep Scale | At baseline and after a 12-week period
  Sleep quality was assessed by Pittsburgh scale, consisting of 19 questions on the perception of oneself and five questions relating to the perception that the roommates of these individuals have about sleep the same. These questions are grouped into seven components, with score of zero to three.
Physical activity levels, evaluated by International Physical Activity Questionnaire (IPAQ) - Long Form. | At baseline and after a 12-week period
  The IPAQ asks about three specific types of activity undertaken in the three domains introduced above and sitting time. The specific types of activity that are assessed are walking, moderate-intensity activities and vigorous intensity activities; frequency (measured in days per week) and duration (time per day) are collected separately for each specific type of activity.

CONTACTS AND LOCATIONS:
Overall Officials: Luiz FM Kruel, phd, Principal Investigator — Federal University of Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No